CLINICAL TRIAL: NCT03713099
Title: A Multicenter Study of the NEUWAVE Flex Microwave Ablation System in the Ablation of Secondary Soft Tissue Lesions of the Lung
Brief Title: NEUWAVE Flexible Probe Study #2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changed study design prior to any patients enrolled.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU_2018_01
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Cancer of the Lung; Lung Cancer; Neoplasms, Lung; Carcinoma, Non-Small Cell Lung; Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma
Keywords: Microwave Ablation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Microwave Ablation (Experimental): Microwave ablations will be performed under general anesthesia via a transbronchial approach performed by an interventional pulmonologist or thoracic surgeon.
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Device: Microwave ablation — Microwave ablations will be performed under general anesthesia via a transbronchial approach by an interventional pulmonologist or thoracic surgeon. Prior to the ablation, the treating physician will perform an endobronchial ultrasound (EBUS) to confirm disease staging.

SUMMARY:
Patients with medically inoperable and operable secondary soft tissue lesion(s) of the lung will have transbronchial microwave ablation performed using cone beam CT for probe guidance and confirmation.

DETAILED DESCRIPTION:
Adult patients with medically inoperable and operable secondary soft tissue lesion(s) of the lung less than 2cm will undergo transbronchial microwave ablation performed by an interventional pulmonologist or thoracic surgeon using cone beam CT imaging for probe guidance and confirmation on ablation outcome. All treated patients will be followed for one year following the ablation procedure for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Patients greater or equal to 18 years of age
3. Performance status 0-2 (Eastern Cooperative Oncology Group classification [ECOG])
4. Willing to fulfill all follow-up visit requirements
5. Medically inoperable and operable secondary soft tissue lesion(s) of the lung
6. A maximum of two ipsilateral soft tissue lesions less than or equal to 2cm in the outer two-thirds of the lung and not closer than 1cm to the pleura. Lesion size must be measured with at least 2-dimensional imaging.

Exclusion Criteria:

1. Scheduled concurrent procedure for the target soft tissue lesion(s) other than those that are lung-related
2. Pregnant or breastfeeding
3. Physical or psychological condition that would impair study participation
4. Patients with uncorrectable coagulopathy at the time of screening
5. Patient with implantable devices, including pacemakers or other electronic implants
6. Prior pneumonectomy or bronchiectasis
7. Severe neuromuscular disease
8. Patient count less than or equal to 50,000/mm cubed
9. ASA (American Society of Anesthesiologists) score of greater than or equal to 4
10. Inability to tolerate anesthesia
11. Expected survival less than 6 months
12. Clinically significant hypertension
13. Chronic, continuous ventilator support, which uses bi-level positive airway pressure (PAP) to improve lung function for severe conditions (however, intermittent PAP, for non-pulmonary conditions, such as sleep apnea, is permitted)
14. Endobronchial soft tissue lesions proximal to the segmental airways
15. Imaging findings of active pulmonary infection
16. The patient was judged unsuitable for study participation by the Investigator for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-31 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Device User Experience Survey | Day of ablation (day 0)
  The Device User Experience Survey is an unvalidated, Sponsor-generated questionnaire aimed to increase the Sponsor's understanding of the usability of the NEUWAVE microwave ablation system. The questionnaire asks approximately 30 questions (includes yes/no responses, rating scales, and fill-in-the-blank sections) and is to be completed by the treating physician at the completion of each ablation. A summary of all treating physician responses will be generated at the completion of the study to summarize the overall user experience with the device.
Technical Success (lesion completely ablated) | Day of ablation (day 0)
  Technical Success is determined by the treating physician and is defined as the ablation zone completely overlapping or encompassing the target lesion plus an ablative margin, as assessed by cone beam CT imaging, immediately following the ablation procedure.
Technique Efficacy (lesion completely ablated) | 30 days post-ablation
  Technique Efficacy is determined by the treating physician and is defined as the ablation zone completely overlapping or encompassing the target lesion plus an ablative margin, as assessed by cone beam CT imaging, at Visit 3 (i.e. 30 days post-ablation).

SECONDARY OUTCOMES:
Adverse Events | 1 year post-ablation
  Any AEs attributable to the ablation procedure, including all device-related, procedure-related, and SAEs, evaluated from the start of the ablation procedure throughout the entirety of the study (i.e. through 1 year post-ablation).
Primary Efficacy Rate | Day of ablation (day 0)
  The Primary Efficacy Rate is the percentage of target lesions successfully eradicated following the first ablation procedure, as assessed using CT imaging by the treating physician on the day of ablation.
Secondary Efficacy Rate | 1 year post-ablation
  The Secondary Efficacy Rate is defined as the percentage of soft tissue lesions that have undergone successful repeat ablations following identification of local soft tissue lesions progression, as assessed using CT imaging by the treating physician throughout the entirety of the study (i.e. 1 year post-ablation).
Target Lesion Recurrence | 1 year post-ablation
  Target Lesion Recurrence is defined as the reappearance of the lesion(s) at the treated site, as assessed using CT imaging by the treating physician throughout the entirety of the study (i.e. through 1 year post-ablation).
Length of Hospital Stay | Day of ablation (day 0)
  The Length of Hospital Stay is defined as the length of time of hospitalization from the end of the ablation procedure to the time of discharge (up to 23 hours post-ablation).
Hospital Readmission Rate | 30 days post-ablation
  The Hospital Readmission Rate is defined as the percentage of patients who were readmitted to the hospital within 30 days of the ablation procedure.

OTHER OUTCOMES:
EORTC QLQ-C30 | 1 year post-ablation
  The EORTC (European Organization for Research and Treatment of Cancer) QLQ-C30 is a quality of life questionnaire with 30 questions aimed specifically for cancer patients. Patients will complete this questionnaire at each study visit.
EORTC QLQ-LC13 | 1 year post-ablation
  The EORTC (European Organization for Research and Treatment of Cancer) QLQ-C30 is a quality of life questionnaire with 13 questions aimed specifically for lung cancer patients. The questionnaire asks patients to rate their responses on a scale from 1-4 (1 being "not at all" and 4 being "very much"). Patients will complete this questionnaire at each study visit.
Numeric Pain Scale | 30 days post-ablation
  The Numeric Pain Scale is a questionnaire where the patient reports their pain on a scale from 0-10 (where 0 is 'no pain' and 10 is 'maximum pain). Patients will complete this questionnaire at each study visit through 30 days post-ablation.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Mayo Clinic, Rochester, Minnesota
  - New York Presbyterian-Weill Cornell Medicine, New York, New York
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Cleveland Clinic, Cleveland, Ohio